CLINICAL TRIAL: NCT05982015
Title: Multicenter, Randomized, Double-blind, Pseudo Treatment-controlled Clinical Study on the Efficacy and Safety of Remote Ischemic Conditioning in Preventing Stroke-associated Pneumonia
Brief Title: Efficacy Study II on Remote Ischemic Conditioning for the Prevention of Stroke-Associated Pneumonia
Acronym: RICA-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RICA-2
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Remote ischemic conditioning (RIC) -200mmHg and best medical management
  Interventions: Device: Remote ischemic conditioning
- Sham group (Sham Comparator): Remote ischemic conditioning (RIC) -60mmHg and best medical management
  Interventions: Device: Sham remote ischemic conditioning

INTERVENTIONS:
Device: Remote ischemic conditioning — The RIC procedure consists of five cycles of unilateral arm ischemia for 5 minutes, which was followed by reperfusion for another 5 minutes. The procedure is performed with an electric, autocontrol device with a cuff that inflated to a pressure of 200 mmHg during the ischemia period. RIC is performed within 24hours after stroke onset, and twice daily for the subsequent 7 days.
  Arms: Intervention group
Device: Sham remote ischemic conditioning — The RIC procedure consists of five cycles of unilateral arm ischemia for 5 minutes, which was followed by reperfusion for another 5 minutes. The procedure is performed with an electric, autocontrol device with a cuff that inflated to a pressure of 60 mmHg during the ischemia period. RIC is performed within 24hours after stroke onset, and twice daily for the subsequent 7 days.
  Arms: Sham group

SUMMARY:
Verifying whether remote ischemic adaptation can reduce the occurrence of stroke related pneumonia in acute stroke patients within 24 hours of onset

DETAILED DESCRIPTION:
Verifying whether remote ischemic adaptation can reduce the occurrence and safety of stroke related pneumonia in acute stroke patients within 24 hours of onset

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old;
* Diagnosis of acute ischemic stroke;
* Remote ischemic conditioning or sham-remote ischemic conditioning can be treated within 24 hours after stroke onset
* NIHSS score≥4;
* Subject or his or her legally authorized representative was able to provide informed consent.

Exclusion Criteria:

* During the screening period, body temperature ≥ 38 ℃;
* Evidence of lung infection, urinary tract infection or other infectious diseases during the screening period
* Expected lifespan less than 7 days
* Mechanical ventilation is expected to be required within 7 days;
* Anti-infective drug were used within 7 days prior to stroke;
* Uncontrolled hypertension with medication (defined as systolic blood pressure ≥200 mmHg and/or diastolic blood pressure ≥110 mmHg);
* There are contraindications for remote ischemic conditioning (such as skin and soft tissue injury, fractures, peripheral arterial disease, etc. in the upper limbs);
* History of autoimmune disease or malignancies;
* Use of immunosuppressive drug within the preceding 3 months;
* Pregnant or lactating, or pregnancy test positive;
* Current participation in another investigational trial;
* Other conditions are not suitable for this trial as evaluated by researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1651 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Stroke-associated pneumonia | 7 days
  Stroke-associated pneumonia incidence rate

SECONDARY OUTCOMES:
Physician diagnosed pneumonia | 7 days
  Physician diagnosed pneumonia incidence rate
Physician diagnosed pneumonia | 8-90 days
  Physician diagnosed pneumonia incidence rate
Modified Rankin scale score from 0 to 1 | 90 days after the onset of symptoms
  In medical and clinical research, the modified Rankin Scale (mRS) is used to assess the degree of disability in patients after a stroke. The scale ranges from 0 to 6, where 0 indicates no symptoms and 6 indicates death.
  On the mRS scale, scores from 0 to 2 usually indicate no or slight disability. Specifically:
  0 points: No symptoms.
  1. point: Symptoms present but no significant disability; able to carry out all usual duties and activities.
  2. points: Slight disability; able to look after own affairs without assistance but unable to carry out all previous activities.
  Therefore, in clinical research, if a treatment or intervention increases the proportion of patients scoring 0 to 1 on the mRS scale, it is generally considered a positive outcome. This means that more patients have a better functional status and lower degree of disability after treatment.
Modified Rankin scale score from 0 to 2 | 90 days
  In medical and clinical research, the modified Rankin Scale (mRS) is used to assess the degree of disability in patients after a stroke. The scale ranges from 0 to 6, where 0 indicates no symptoms and 6 indicates death.
  On the mRS scale, scores from 0 to 2 usually indicate no or slight disability. Specifically:
  0 points: No symptoms.
  1. point: Symptoms present but no significant disability; able to carry out all usual duties and activities.
  2. points: Slight disability; able to look after own affairs without assistance but unable to carry out all previous activities.
  Therefore, in clinical research, if a treatment or intervention increases the proportion of patients scoring 0 to 2 on the mRS scale, it is generally considered a positive outcome. This means that more patients have a better functional status and lower degree of disability after treatment.
Modified Rankin scale scores | 90 days
  Shift analysis. In medical and clinical research, the modified Rankin Scale (mRS) is used to assess the degree of disability in patients after a stroke. The scale ranges from 0 to 6, where 0 indicates no symptoms and 6 indicates death.
  On the mRS scale, scores from 0 to 2 usually indicate no or slight disability. Specifically:
  0 points: No symptoms.
  1. point: Symptoms present but no significant disability; able to carry out all usual duties and activities.
  2. points: Slight disability; able to look after own affairs without assistance but unable to carry out all previous activities.
  Therefore, in clinical research, if a treatment or intervention increases the proportion of patients scoring 0 to 2 on the mRS scale, it is generally considered a positive outcome. This means that more patients have a better functional status and lower degree of disability after treatment.
EQ-5D-5L scores | 90 days
  The scores of EQ-5D-5L. The five dimensions included in EQ-5D-5L are:
  Mobility: This dimension assesses the person's ability to walk about. Self-Care: This evaluates the individual's ability to wash or dress themselves. Usual Activities: This covers work, study, housework, family or leisure activities.
  Pain/Discomfort: This measures the level of pain or discomfort experienced by the individual.
  Anxiety/Depression: This assesses the person's psychological state, in terms of levels of anxiety or depression.
  Each of these five dimensions has five levels of severity:
  Level 1: No problems Level 2: Slight problems Level 3: Moderate problems Level 4: Severe problems Level 5: Extreme problems
NIHSS stroke scale scores | 24 hours
  The scores of NIHSS stroke scale. The total NIHSS score can range from 0 to 42, with:
  0: Indicating no stroke symptoms. 1-4: Indicating a minor stroke. 5-15: Indicating a moderate stroke. 16-20: Indicating a moderate to severe stroke. 21-42: Indicating a severe stroke. The NIHSS is useful in evaluating the effect of acute stroke treatments, predicting patient outcomes, and assessing the progression of stroke symptoms.
NIHSS stroke scale scores | 7 days
  The scores of NIHSS stroke scale. The total NIHSS score can range from 0 to 42, with:
  0: Indicating no stroke symptoms. 1-4: Indicating a minor stroke. 5-15: Indicating a moderate stroke. 16-20: Indicating a moderate to severe stroke. 21-42: Indicating a severe stroke. The NIHSS is useful in evaluating the effect of acute stroke treatments, predicting patient outcomes, and assessing the progression of stroke symptoms.
Urinary tract infections | 7 days
  Urinary tract infections incidence rate
Infections | 7 days
  Infections incidence rate
All-cause mortality | 90 days
  All-cause mortality incidence rate
Inpatient days | 90 days
  Total inpatient days

OTHER OUTCOMES:
Spots of skin bleeding within 7 days | 7 days
  Number of subjects who have skin bleeding points within 7 days
Red or swollen arms within 7 days | 7 days
  Number of subjects who have red or swollen arms within 7 days
Dizziness within 7 days | 7 days
  Number of subjects who have dizziness within 7 days
Nausea within 7 days | 7 days
  Number of subjects who have nausea within 7 days
Palpitations within 7 days. | 7 days
  Number of subjects who have palpitations within 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Chuanjie Wu, M.D., Study Director — Xuanwu Hospital of Capital Medical University
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Background] Westendorp WF, Vermeij JD, Zock E, Hooijenga IJ, Kruyt ND, Bosboom HJ, Kwa VI, Weisfelt M, Remmers MJ, ten Houten R, Schreuder AH, Vermeer SE, van Dijk EJ, Dippel DW, Dijkgraaf MG, Spanjaard L, Vermeulen M, van der Poll T, Prins JM, Vermeij FH, Roos YB, Kleyweg RP, Kerkhoff H, Brouwer MC, Zwinderman AH, van de Beek D, Nederkoorn PJ; PASS investigators. The Preventive Antibiotics in Stroke Study (PASS): a pragmatic randomised open-label masked endpoint clinical trial. Lancet. 2015 Apr 18;385(9977):1519-26. doi: 10.1016/S0140-6736(14)62456-9. Epub 2015 Jan 20. PMID 25612858
- [Background] Kalra L, Irshad S, Hodsoll J, Simpson M, Gulliford M, Smithard D, Patel A, Rebollo-Mesa I; STROKE-INF Investigators. Prophylactic antibiotics after acute stroke for reducing pneumonia in patients with dysphagia (STROKE-INF): a prospective, cluster-randomised, open-label, masked endpoint, controlled clinical trial. Lancet. 2015 Nov 7;386(10006):1835-44. doi: 10.1016/S0140-6736(15)00126-9. Epub 2015 Sep 3. PMID 26343840
- [Background] Hoffmann S, Harms H, Ulm L, Nabavi DG, Mackert BM, Schmehl I, Jungehulsing GJ, Montaner J, Bustamante A, Hermans M, Hamilton F, Gohler J, Malzahn U, Malsch C, Heuschmann PU, Meisel C, Meisel A; PREDICT Investigators. Stroke-induced immunodepression and dysphagia independently predict stroke-associated pneumonia - The PREDICT study. J Cereb Blood Flow Metab. 2017 Dec;37(12):3671-3682. doi: 10.1177/0271678X16671964. Epub 2016 Oct 14. PMID 27733675
- [Background] Chamorro A, Meisel A, Planas AM, Urra X, van de Beek D, Veltkamp R. The immunology of acute stroke. Nat Rev Neurol. 2012 Jun 5;8(7):401-10. doi: 10.1038/nrneurol.2012.98. PMID 22664787
- [Background] Iadecola C, Anrather J. The immunology of stroke: from mechanisms to translation. Nat Med. 2011 Jul 7;17(7):796-808. doi: 10.1038/nm.2399. PMID 21738161
- [Background] Chamorro A, Urra X, Planas AM. Infection after acute ischemic stroke: a manifestation of brain-induced immunodepression. Stroke. 2007 Mar;38(3):1097-103. doi: 10.1161/01.STR.0000258346.68966.9d. Epub 2007 Jan 25. PMID 17255542
- [Background] Randhawa PK, Bali A, Jaggi AS. RIPC for multiorgan salvage in clinical settings: evolution of concept, evidences and mechanisms. Eur J Pharmacol. 2015 Jan 5;746:317-32. doi: 10.1016/j.ejphar.2014.08.016. Epub 2014 Aug 28. PMID 25176179
- [Derived] Jia L, Hou C, Mei Q, Zhang B, Zhao W, Zhao H, Shang S, Guo X, Ma Q, Song H, Li C, Meng R, Xu W, Wang Y, Xu G, Wu C, Ji X, Investigators FTR. Remote ischemic conditioning for the prevention of stroke-associated pneumonia (RICA-2): protocol for a multicenter, prospective, randomized, double-blind, sham-controlled phase III trial. Trials. 2025 Oct 16;26(1):419. doi: 10.1186/s13063-025-09140-x. PMID 41102804